CLINICAL TRIAL: NCT02568670
Title: Removal Peripheral Intravenous Catheters According to Clinical Signs or Every 96 Hours: A Non Inferiority Study (ResPeCt)
Brief Title: Removal Peripheral Intravenous Catheters According to Clinical Signs or Every 96 Hours: A Non Inferiority Study
Acronym: ResPeCt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Patricia Vendramim, MsC, PhD student, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15849513.2.0000.5487
Record Dates: First submitted 2015-09-21; First posted 2015-10-06 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Phlebitis
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- according to clinical signs (Experimental): removal the peripheral catheter according to clinical signs
  Interventions: Other: clinical signs
- sistematically every 96 hours (No Intervention): removal the peripheral catheter every 96 hours

INTERVENTIONS:
Other: clinical signs — to remove the peripheral venous catheter according clinical signs
  Arms: according to clinical signs

SUMMARY:
This is a two-centers, open label, prospective, randomized, noninferiority controlled trial with cost-effectiveness analysis to verify if is non inferior to remove peripheral intravenous catheter according to clinical signs in relation to every 96 hours.

DETAILED DESCRIPTION:
The care practice standards related to infusion therapy (IT) are stipulated and regulated by US institutions, such as the Infusion Nurses Society (INS) and the Center for Disease and Control (CDC), and, in Brazil, by the Brazilian National Health Surveillance Agency (ANVISA). Within this topic, the investigators can mention peripherally administered IT through peripheral intravenous catheters (PIC) as the most used one, since this is less complex and less invasive, and it offers a lower risk of severe complications compared to central line IT.

PIC placement, maintenance and removal procedures are not free of complications, and in order to prevent them, regulatory agencies publish formal recommendations. One of these refers to the time the PIC remains at the same site (residence time), which has been determined to be 96 hours for the adult population, i.e., it should be removed and punctured again at another site, systematically, even if not showing any inflammatory sign within 96 hours.

Following literature review, one can see that these recommendations are based on limited evidence, and supported by data from old studies. For this reason, the investigators discuss if employing a systematic and elective change procedure for adults would be the best option, as the investigators have taken some aspects into consideration, such as: Patient safety - The PIC dwell time at the placement site, as shown by research results, has increased throughout the decades to 24, 48, 72, and 96 hours. If the PIC change is performed on a child who, theoretically, is a less immune-competent patient as compared to adults, this is performed according to clinical signs, then the investigators can conclude that adopting the same procedure for adults would be safe. Peripheral venous depletion - Logic leads us to consider that the less the investigators puncture a patient, more access is available, and less outcomes with IT-specific complications occur. Patient satisfaction - With reduced exposures to painful and invasive events, the patient will also benefit from it. Few patients refrain from showing dissatisfaction when the PIC is to be placed again electively. Quality - Producing scientific evidence and adopting the best practices in hospital environments is practicing quality. Economic aspects - If these PIC changes were less frequent, they would necessarily imply less spending with inputs and devices, as well as less time spent by the team performing the procedure, which represents less cost and workload. Occupational safety - Studies show an estimated relationship between the occurrence of an accident with biological material and performing invasive procedures. Reducing the number of punctures performed by a professional, in addition to decreasing the workload, may reduce the exposure to risk and accidents.

Research studies carried out mostly in Australia aim at showing that the systematic PIC removal and change do not bring benefits, when compared to change based on clinical manifestations. However, a systematic review study in 2010 did not find conclusive evidence, and suggested the development of other projects in several regions, of different natures and realities, so as to further mature the hypothesis. To support this, the INS has also formally stated that this theme is a research priority at this time.

ELIGIBILITY:
Inclusion Criteria:

* any medical diagnosis, except for those stated as exclusion criteria, and
* with a therapeutic proposal of undergoing the therapy for at least 96 hours, or four days;
* agree with the proposals expressed in the Informed Consent Form (ICF); and
* have a catheter that has not been placed at the ER.

Exclusion Criteria:

* medical diagnosis of immunosuppression or receiving immunosuppressants;
* using more than one peripheral catheter simultaneously;
* refusing to take part in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1305 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
presence of phlebitis | from catheter fixation, during the indwell time of the catheter, until the removal of it. For the control group, it will be up to 96 hours. From the interventional group, there is no time predict, average five or six days
  phlebitis (phlebitis/1000 peripheral venous catheters-day), stratified by severity.

SECONDARY OUTCOMES:
presence of other complications related peripheral intravenous (PIC) therapy in the two groups | from catheter fixation, during the indwell time of the catheter, until the removal of it. For the control group, it will be up to 96 hours. From the interventional group, there is no time predict, average five or six days
  complications (event/1000 peripheral venous catheters-day)
time interval for peripheral intravenous catheter (PIC) changes | For the control group, it will be up to 96 hours. From the interventional group, there is no time predict, average five or six days
  Through these measures:
  * length of stay in hours / avp-day * 1000
  * length of stay in hours / patient
  From catheter fixation, during the indwell time of the catheter, until the removal of it.
total number of peripheral intravenous catheter (PIC) | After randomization, from the first venous puncture, catheter fixation, until the removal of it, during the hospitalization. Average six days
  Total number of peripheral intravenous catheter (PIC) used in the two groups. Through these measures:
  * number of PIC re-inserted / patient
  * number of PIC re-inserted / avp-day * 1000
  * number of venous punctures to obtain access / patient
Cost | during the hospitalization, in average 5 to 6 days
  . Cost of 30 minutes of professional time for peripheral intravenous puncturing (PIP).
  * Cost of inputs for each insertion - soap for cleaning, examination gloves, pre-filled syringe with saline, alcohol swab, PIC, intermediate type extension y, two valve connectors, fixture and transparent semi-permeable membrane covering polyurethane.
  * Cost 10 minutes from time professional (practical nurse) for removal.
  * Cost of inputs to remove the PIC - alcohol swab and anti-hemorrhagic coverage.
  * Cost of daily patient hospitalization related to the catheter dwell time.
The experience of the patient | the questionnaire will be applied at the time of hospital discharge, hospitalization with average 6 days
  applying a questionnaire of assessment of the experience of the patient in use of peripheral venous catheter at the end of admission, wich was elaborated by the author and validated by expert judges. Principal contents: Information and education: guidance on research and care given peripheral IT Physical comfort: pain or discomfort procedures Emotional support: considered in this study as trust / security transmitted and perceived Respect for patient preferences: flexibility to accept small patient preferences Involvement of family and friends: identify the participation of people significant to patient and allow shared decision Continuity and transition: if care is independent continuous service location within the institution General impressions: courtesy and availability of staff Overall satisfaction: at the end the experience was satisfying Complaints: originated by dissatisfaction reasons Fidelity: creation of the trust, return and referral to another service

CONTACTS AND LOCATIONS:
Locations (1):
- Samaritano Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Vendramim P, Avelar AFM, Rickard CM, Pedreira MDLG. The RESPECT trial-Replacement of peripheral intravenous catheters according to clinical reasons or every 96 hours: A randomized, controlled, non-inferiority trial. Int J Nurs Stud. 2020 Jul;107:103504. doi: 10.1016/j.ijnurstu.2019.103504. Epub 2020 Jan 11. PMID 32334176